CLINICAL TRIAL: NCT03453996
Title: Evaluating Enhanced Clinical Decision Support for Prevention of Contrast-Induced Acute Kidney Injury in Cardiac Catheterization
Brief Title: Contrast RISK (Reducing Injury Sustained by Kidneys)
Acronym: Contrast RISK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REB17-0039
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2021-05

CONDITIONS: Acute Kidney Injury (Nontraumatic); Coronary Artery Disease
Keywords: acute kidney injury; heart disease; cardiac catheterization
MeSH Terms: conditions — Acute Kidney Injury; Coronary Artery Disease; Heart Diseases | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cardiologists will receive computerized clinical decision support information for CI-AKI prevention for patients identified above the median (> 5%) risk of AKI based on the NCDR risk prediction model for CI-AKI.
  Interventions: Other: Intervention
- Control (Other): Usual care.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Computerized clinical decision support intervention. This intervention consists of 2 decision support components for CI-AKI prevention:
  1. Estimation of safe contrast limit to reduce the relative risk of CI-AKI by 20% (ePRISM Acute Kidney Injury Model with Contrast Sensitivities and Dialysis Risk software from Health Outcomes Sciences)
  2. Patient weight and left ventricular end diastolic pressure (LVEDP) based intravenous crystalloid fluid recommendation.
  Arms: Intervention
Other: Control — Usual procedural care provided by cardiologist without introduction of the computerized clinical decision support information.
  Arms: Control

SUMMARY:
Diagnostic and therapeutic cardiac catheterization procedures are important interventions to reduce the risk of death, avoid future cardiovascular events, and improve quality of life of people with heart disease. However, exposure to the radiocontrast dyes required for these procedures can lead to contrast-induced acute kidney injury (CI-AKI); a common and costly complication. There are accurate ways to identify patients at increased risk of this complication and strategies to prevent CI-AKI. This involves ensuring that patients who are at risk have procedures done with the minimum amount of X-ray contrast dye required, and that they receive optimal intravenous fluids at the time of the procedure.

This study will evaluate the implementation of a strategy where computerized decision support tools are used to help doctors identify patients at risk of CI-AKI, as well as make decisions about how much contrast dye to use and how much intravenous fluid to provide to patients who are identified at risk of CI-AKI in cardiac catheterization.

DETAILED DESCRIPTION:
Overview: Randomized stepped-wedge trial to evaluate the impact of implementing a computerized decision support strategy that incorporates CI-AKI risk prediction and calculation of safe contrast dye limits and intravenous fluid recommendations.

Study Population: Adult patients undergoing diagnostic or interventional coronary angiography procedures will be eligible if not already receiving dialysis. Patients receiving emergency primary percutaneous coronary intervention (PCI) for ST-elevation myocardial infarction will be excluded.

Intervention: Multivariable clinical risk prediction model to estimate risk of CI-AKI and safe contrast limits for patients above the median (>5%) predicted risk of CI-AKI. Intravenous fluids recommendations based on weight and left-ventricular end-diastolic pressure will also be provided for patients identified above the median risk of CI-AKI.

The National Cardiovascular Data Registry (NCDR) Cath-PCI Registry AKI risk model will be used to estimated the predicted risk of CI-AKI, and safe contrast limits will be estimated using the ePRISM, Acute Kidney Injury Model with Contrast Sensitivities and Dialysis Risk (Health Outcomes Sciences) software, incorporated within the Alberta Provincial Project for Outcomes Assessment in Coronary Heart Disease (APPROACH) Cardiac Catheterization software.

Study Design: Using a stepped-wedge design, clusters of cardiologists who perform diagnostic or therapeutic cardiac catheterization in each centre will be randomized to be introduced to the intervention at sequential time points spaced over 20 months. At each step, cardiologists who have not yet been randomized will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing diagnostic coronary angiography or coronary intervention in Alberta

Exclusion Criteria:

* Emergency primary percutaneous coronary intervention for ST-elevation myocardial infarction
* Receiving dialysis at time of cardiac catheterization procedure
* Non-Alberta resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7280 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 4 days after procedure
  >26 micromol/L or 50% increase in serum creatinine

SECONDARY OUTCOMES:
Post-Procedural Hospital Bed Days | Thirty days after procedure
  Number of days in hospital including length of stay plus readmissions up to 30 days after procedure
Death | One year after procedure
  Total mortality
Change in eGFR | One year after procedure
  Change in eGFR at one year fro pre-procedural baseline (estimated using CKD-EPI equation)
Cardiac Events | One year after procedure
  Hospital admission for angina, myocardial infarction, heart failure, or unplanned revascularization procedure (excluding staged procedures)
Kidney Events | On year after procedure
  Hospital admission for acute kidney injury or dialysis
End-stage Kidney Disease | One year after procedure
  Kidney failure requiring dialysis, kidney transplantation, or conservative management of kidney failure with eGFR<15 mL/min/1.73m2
Generic Quality of Life | One year after procedure
  EQ-5D
Cardiovascular-specific quality of life | One year after procedure
  Seattle Angina Questionnaire
Contrast Volume | Day of procedure
  Volume of contrast used for each case
Intravenous Fluid | Day of procedure
  Volume of intravenous fluids used for each case

OTHER OUTCOMES:
Total direct health care costs | One year after procedure
  Total direct health care costs
Cost per quality-adjusted life year | One year after procedure
  Total direct health care costs per quality adjusted life year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T James, MD PhD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
Due to Alberta privacy regulations, unable to share data

REFERENCES:
- [Background] Tsai TT, Patel UD, Chang TI, Kennedy KF, Masoudi FA, Matheny ME, Kosiborod M, Amin AP, Weintraub WS, Curtis JP, Messenger JC, Rumsfeld JS, Spertus JA. Validated contemporary risk model of acute kidney injury in patients undergoing percutaneous coronary interventions: insights from the National Cardiovascular Data Registry Cath-PCI Registry. J Am Heart Assoc. 2014 Dec;3(6):e001380. doi: 10.1161/JAHA.114.001380. PMID 25516439
- [Background] Amin AP, Bach RG, Caruso ML, Kennedy KF, Spertus JA. Association of Variation in Contrast Volume With Acute Kidney Injury in Patients Undergoing Percutaneous Coronary Intervention. JAMA Cardiol. 2017 Sep 1;2(9):1007-1012. doi: 10.1001/jamacardio.2017.2156. PMID 28678988
- [Background] Allen DW, Ma B, Leung KC, Graham MM, Pannu N, Traboulsi M, Goodhart D, Knudtson ML, James MT. Risk Prediction Models for Contrast-Induced Acute Kidney Injury Accompanying Cardiac Catheterization: Systematic Review and Meta-analysis. Can J Cardiol. 2017 Jun;33(6):724-736. doi: 10.1016/j.cjca.2017.01.018. Epub 2017 Feb 1. PMID 28545621
- [Derived] James MT, Har BJ, Tyrrell BD, Faris PD, Tan Z, Spertus JA, Wilton SB, Ghali WA, Knudtson ML, Sajobi TT, Pannu NI, Klarenbach SW, Graham MM. Effect of Clinical Decision Support With Audit and Feedback on Prevention of Acute Kidney Injury in Patients Undergoing Coronary Angiography: A Randomized Clinical Trial. JAMA. 2022 Sep 6;328(9):839-849. doi: 10.1001/jama.2022.13382. PMID 36066520
- [Derived] James MT, Har BJ, Tyrrell BD, Ma B, Faris P, Sajobi TT, Allen DW, Spertus JA, Wilton SB, Pannu N, Klarenbach SW, Graham MM. Clinical Decision Support to Reduce Contrast-Induced Kidney Injury During Cardiac Catheterization: Design of a Randomized Stepped-Wedge Trial. Can J Cardiol. 2019 Sep;35(9):1124-1133. doi: 10.1016/j.cjca.2019.06.002. Epub 2019 Jun 7. PMID 31472811
- See also: Health Outcomes Sciences — http://www.h-outcomes.com/
- See also: Alberta Provincial Project for Outcomes Assessment in Coronary Heart Disease — http://www.approach.org/